CLINICAL TRIAL: NCT00170287
Title: Substrate Modification Study in Patients Getting an ICD
Brief Title: SMS: Substrate Modification Study in Patients Getting an Implantable Cardioverter Defibrillator (ICD)
Acronym: SMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEN_G_CA_3
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2017-09

CONDITIONS: Tachycardia, Ventricular
Keywords: Unstable Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ICD Therapy plus VT-Ablation
  Interventions: Procedure: ICD Ablation plus VT-ablation
- 2 (Active Comparator): ICD Therapy only
  Interventions: Device: ICD Therapy

INTERVENTIONS:
Procedure: ICD Ablation plus VT-ablation — ICD-Therapy for the treatment of unstable VT´s plus catheter ablation for substrate modification
  Arms: 1
Device: ICD Therapy — ICD Therapy for the Treatment of unstable VT´s
  Arms: 2

SUMMARY:
The present standard of care for the management of unstable ventricular tachycardia (VT) in the setting of chronic coronary artery disease is the placement of an implantable cardioverter defibrillator (ICD) after the initial episode, and radiofrequency ablation and/or antiarrhythmic medication in the event of recurrences causing frequent ICD interventions.

The primary purpose of this randomized study is the assessment of recurrences of unstable VT in patients who undergo ICD implantation plus substrate ablation after the initial episode compared to patients who only undergo ICD implantation. Thus the primary purpose is an improvement in the quality of life. A decrease in mortality is not a primary purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease documented by coronary angiography. For the purpose of this study, coronary artery disease will be defined as the presence of a 50% or more diameter stenosis of the left main or of a 75% or more diameter stenosis of the left anterior descending, circumflex or right coronary arteries, or the history of a surgical or percutaneous revascularization procedure.
* Left ventricular ejection fraction < 40% as estimated by echocardiography or contrast ventriculography within the previous 30 days.
* Clinical unstable VT without reversible factors (acute ischemia or antiarrhythmic medications as defined below). Unstable VT can have one of the following clinical presentations:

  * Hypotensive VT without major neurologic dysfunction;
  * Syncope; or
  * Cardiac arrest.

Exclusion Criteria:

* Age < 18 years or > 80 years
* Protruding left ventricular (LV) thrombus on pre-ablation echocardiogram
* Acute myocardial infarction within the preceding 2 months
* Class IV New York Heart Association (NYHA) heart failure
* Valvular heart disease or mechanical heart valve precluding access to the left ventricle
* Unstable angina
* Cardiac surgery within the past 2 months
* Serum creatinine > 220 mmol/L (2.5 mg/dL)
* Thrombocytopenia or coagulopathy
* Contraindication to heparin
* Pregnancy
* Acute illness or active systemic infection
* Other disease process likely to limit survival to less than 12 months
* Significant medical problem that, in the opinion of the principal investigator, would preclude enrollment into the study
* Participation in another investigational study
* Unwillingness to participate or lack of availability for follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2002-05; Primary Completion 2010-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Time to the first documented recurrence of any sustained VT/ventricular fibrillation (VF) during the follow-up period | 12 Months

SECONDARY OUTCOMES:
All appropriate ICD therapies (number of shocks, number of antitachycardia pacing therapies) | 12 Months
Quality of life | 12 Months
Number of hospital readmissions due to a cardiac indication | 12 Months
Severe clinical events | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, MD, Principal Investigator — Allgemeines Krankenhaus St. Georg
Locations (7):
- Skejby Skygehus, Aarhus, Denmark
- Germany (6):
  - Herz- und Gefäßklinik GmbH, Bad Neustadt / Saale
  - Berufsgenossenschaftliche Kliniken Bergmannsheil, Bochum
  - Klinikum der J.W. Goethe Universität, Frankfurt
  - Allgemeines Krankenhaus St. Georg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuck KH, Tilz RR, Deneke T, Hoffmann BA, Ventura R, Hansen PS, Zarse M, Hohnloser SH, Kautzner J, Willems S; SMS Investigators. Impact of Substrate Modification by Catheter Ablation on Implantable Cardioverter-Defibrillator Interventions in Patients With Unstable Ventricular Arrhythmias and Coronary Artery Disease: Results From the Multicenter Randomized Controlled SMS (Substrate Modification Study). Circ Arrhythm Electrophysiol. 2017 Mar;10(3):e004422. doi: 10.1161/CIRCEP.116.004422. PMID 28292751